CLINICAL TRIAL: NCT05651022
Title: A Phase 1/2, Open-Label, Multi-Center, Dose Escalation and Expansion Study Evaluating the Safety, Tolerability and Clinical Activity of DECOY20 as Monotherapy and in Combination With Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: Study of DECOY20 With or Without Tislelizumab in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indaptus Therapeutics, Inc (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INDP-D101
Record Dates: First submitted 2022-11-18; First posted 2022-12-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult; HCC - Hepatocellular Carcinoma; CRC (Colorectal Cancer); Pancreatic Adenocarcinoma; NSCLC Non-small Cell Lung Cancer; Squamous Cell Cancer of the Head and Neck; UC (Urothelial Cancer); MSI-H Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: Subjects received a single dose of Decoy20 at one of two assigned dose levels on Week 1 Day 1. Subjects were observed for 28 days for dose-limiting toxicity in the single ascending dose Part 1. Subjects enrolled in Part 2a and 2b receive continuous weekly doses of Decoy20 as monotherapy at the dose(s) determined from Part 1. Subjects enrolled in Part 2c will receive continuous weekly doses of Decoy20 at the dose(s) determined from Part 2a in combination with tislelizumab at its approved dose and schedule.
  Safety and preliminary anti-tumor activity will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): A single dose of Decoy20 at a dose of 3 x 10^7 KB or 7 x 10^7 KB
  Interventions: Drug: Decoy20
- Parts 2a and 2b (Experimental): Decoy20 administered weekly at a dose of 3 x 10^7 KB or 7 x 10^7 KB
  Interventions: Drug: Decoy20
- Part 2c (Experimental): Decoy20 administered weekly at either 3 x 10^7 KB or 7 x 10^7 KB. Both will be administered with tislelizumab at 200mg Q3W.
  Interventions: Drug: Decoy20; Drug: Tislelizumab

INTERVENTIONS:
Drug: Decoy20 — Decoy20 is a novel, systemically administered multiple Toll-like receptor (TLR) agonist-based cancer immunotherapy.
Drug: Tislelizumab — Tislelizumab is a PD-1 inhibitor.
  Arms: Part 2c

SUMMARY:
INDP-D101 is a Phase 1/2, open-label, multi-center, dose escalation and expansion study evaluating the safety, tolerability and clinical activity of Decoy20 as monotherapy and in combination with tislelizumab in patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Decoy20, is a novel, systemically administered multiple Toll-like receptor (TLR) agonist-based cancer immunotherapy.

INDP-D101 is a Phase 1/2, open-label, multi-center, 3+3 dose escalation and expansion study evaluating the safety, tolerability and clinical activity of Decoy20 in subjects with advanced solid tumors. The study will include 2 parts:

In Part 1, Subjects will receive a single dose of Decoy20 at one of up to three assigned dose levels on Week 1 Day 1 (SAD). Subjects will be observed for 28 days for dose limiting toxicity. Safety will be assessed by a safety review committee (SRC), comprised of investigators and the study sponsor, and subsequently will recommend the dose of Decoy20 to take forward.

Part 2 began when a single dose recommended from Part 1 was identified to confirm the safety of weekly administration of Decoy20 in approximately 54 to 90 subjects. More than one dose may be studied in Part 2 that is at or below the MTD determined in Part 1. Eligible subjects must have one of the following locally advanced or metastatic tumor types: hepatocellular carcinoma (HCC), colorectal cancer (CRC) with liver metastasis, urothelial cancer, squamous cell carcinoma of the head and neck (SCCHN), adenocarcinoma of the pancreas, non-small cell lung cancer (NSCLC). Part 2 is further divided into 3 parts a Safety Run-In (Part 2a), a Dose Expansion (Part 2b) and a Combination with a PD-1 inhibitor, tislelizumab (Part 2c).

Part 2a enrolls 6 subjects in a staggered manner, and each subject receives 4 weekly doses of Decoy20 identified in Part 1. Safety data for each of these subjects is collected for 4 weeks after the subjects' 4th Decoy20 dose for acute and delayed toxicity. This data is reviewed by the SRC and a determination of one or more tolerable doses of Decoy20 for Part 2b is made.

Part 2b further evaluates and confirms the safety and preliminary efficacy of continuous weekly Decoy20 administration for up to 1 year. The SRC continues to meet and reviews data on an ongoing or ad-hoc basis during Part 2b of the study to ensure that there are no undue risks to study subjects and to confirm one or more tolerable doses for Phase 2.

Part 2c will evaluate the safety and tolerability of Decoy20 in combination with tislelizumab. The SRC will continue to meet and review data on an ongoing or ad-hoc basis during Part 2c of the study to ensure that there are no undue risks to study subjects and to confirm one or more tolerable Phase 2 doses and sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 years or older.
2. Histologically confirmed diagnosis of locally advanced or metastatic solid tumor. For Part 2, subjects must have one of the following locally advanced or metastatic tumor types: hepatocellular carcinoma (HCC), colorectal cancer (CRC) with liver metastasis, urothelial cancer, squamous cell carcinoma of the head and neck (SCCHN), adenocarcinoma of the pancreas, non-small cell lung cancer (NSCLC), dMMR/MSI-High tumor (Part 2c only).
3. Subject must have exhausted all available therapy or have declined treatment or treatment is contraindicated. Subjects with tumors that have known actionable molecular alteration such as EGFR, ALK, ROS-1, BRAF, RET, MET, and KRAS must have progressed on directed molecular therapy. For Part 2c, participants with a tumor type for which a CPI has been approved must have received a CPI during one or more lines of therapy.
4. Measurable disease (at least 1 measurable lesion) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as defined by tumor type.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy of at least 3 months.
7. Female subjects must be of non-childbearing potential (surgically sterile or at least 2 years postmenopausal) or agree to use a highly effective contraception method while receiving treatment with Decoy20 and for 30 days after the last dose of Decoy20.
8. Male subjects must utilize reliable contraceptive precautions for the duration of Decoy20 treatment and 30 days after the last dose of Decoy20.
9. Adequate organ function as demonstrated by baseline laboratory assessment.
10. Left ventricular ejection fraction (LVEF) ≥ 45% by echocardiogram (ECHO) or multi-gated acquisition scan (MUGA).
11. Recovered from toxicities due to prior therapies.
12. Willing and able to comply with all scheduled visits, laboratory tests, and other study procedures including mandatory pre-treatment and on- treatment biopsies for subjects enrolled to Part2.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Has an active systemic (viral, bacterial, or fungal) infection or requiring treatment.
3. Received radiotherapy within 28 days of the first dose of Decoy20. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
4. Received prior chemotherapy, targeted therapy or immunotherapy within 28 days or 5 half-lives from W1D1, whichever is shorter.
5. Received systemic corticosteroid therapy > 5 mg/day of prednisone or equivalent dose of another corticosteroid within 1 week or 5 half-lives (whichever is shorter) from the start of study drug or is expected to require it during the course of the study (topical and inhaled steroids are permitted).
6. Has radiographically detected primary central nervous system (CNS) metastases or symptomatic CNS involvement (including leptomeningeal carcinomatosis, cranial neuropathies or mass lesions that cause spinal cord compression). Participants with brain metastases (either treated or deemed unnecessary to treat) that have been stable by neuroimaging for at least 4 weeks will be eligible.
7. Clinical evidence of significant coagulopathy during Screening (e.g., deep vein thrombosis or pulmonary embolism) or history of significant uncontrolled coagulopathy (participants with HCC must have prothrombin time (PT) < 4 seconds above ULN or international normalized ratio [INR] < 1.7) or participants with diagnosis of a new thrombotic event within 90 days prior to Decoy20 dosing.
8. Has an active secondary malignancy in addition to the primary, excluding low-risk neoplasms as determined by the Investigator (e.g., non-metastatic basal cell or squamous cell skin carcinoma) and other indolent malignancies will be allowed after discussion with the Sponsor).
9. Has a history of or active infection with HIV 1 or 2, a history of or active infection with HBV based upon HBV antigenemia or viral load, or positive read for hepatitis C virus ([HCV] viral load >15 IU/mL) at Screening. 10. Has a history of known genetic predisposition to HLH/MAS.

11. Has undergone splenectomy, has an active chronic liver disease, Wilson's disease, hemochromatosis, primary biliary cirrhosis, primary sclerosing cholangitis, genetic hemochromatosis, history of or planned liver transplant for end-stage liver disease of any etiology, documented history of advanced liver fibrosis or history of cirrhosis and/or hepatic decompensation including ascites requiring paracentesis rather than medical therapy, modified Child-Pugh B or C, clinically relevant hepatic encephalopathy within the preceding 6 months, or variceal bleeding. 12. Has received a vaccine within 14 days of W1D1 13. Has active autoimmune disease. 14. Has a history of significant CNS disease, such as stroke (past history of transient ischemic attacks more than 3 months ago and controlled is allowed) or uncontrolled and unstable epilepsy. 15. Has severe pulmonary interstitial disease and/or oxygen saturation on room air < 92%. 16. Baseline Q-T correlated (QTc) interval of > 470 msec for females and > 450 msec for males calculated using Fridericia's formula. 17. New York Heart Association Class III or IV cardiac disease, or myocardial ischemia or infarction within 180 days of Screening, vaso-vagal sensitivity, unstable angina, coronary/peripheral artery bypass graft, worsening/ decompensated heart failure within the past 6 months, or any other clinically significant cardiac abnormality that, in the judgement of the Investigator, would pose a health risk to the subject. 18. Major surgical procedure within 4 weeks prior to first dose of Decoy20, or anticipation of need for a major surgical procedure, during the study. 19. Any other acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or Decoy20 administration. 20. Has received investigational therapy within 28 days or 5 half-lives of the start of study drug. 21. Unwillingness or inability to comply with procedures required in this protocol. 22. Known allergy or hypersensitivity to Decoy20 or one of the ingredients of Decoy20. 23. For Part 2c, participants with ongoing immune-related adverse events (irAEs) from other agents or who required permanent discontinuation of prior ICIs due to irAEs. Participants with a prior history of Grade 3 or higher irAE except for those with a history of an immune-related endocrinopathy which is currently treated and clinically stable. Participants with a history of (non-infectious) Grade 2 or higher pneumonitis that required steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with dose-limiting toxicities (DLTs) | Through study completion, up to 3 years
  A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medication. The relatedness and severity of treatment emergent adverse events will utilize the National Cancer Institute Common Toxicity Criteria for adverse events (NCI-CTCAE) for assessment.
Percentage of subjects with Adverse Events (AEs) | Through completion, up to 3 years
  The count and percentage of subjects with AEs and Treatment Emergent Adverse Events (TEAEs) will be assessed for all subjects.
Maximum Tolerated Dose (MTD) of Decoy20 | Up to 2 years
  The MTD is defined as the highest dose level at which no more than 1 out of 6 subjects experiences Dose Limiting Toxicity during the first 28 days after dosing of Decoy20.
Recommended Phase 2 Dose (RP2D) of Decoy20 | Up to 2.5 years
  The highest dose level that is declared to be safe and tolerable by the investigators and the sponsor.

SECONDARY OUTCOMES:
Anti-Drug Antibodies (ADA) | Up to 3 years
  The incidence of ADAs will be assessed.
Neutralizing Antibodies (NAbs) | Up to 3 years
  The incidence of antibodies neutralizing Decoy20 will be assessed
Maximum drug concentration (Cmax) of Decoy20 | Up to 3 years
  The blood pharmacokinetic parameter, Cmax, will be assessed pre-dose and up to 28 days post-dose after administration of Decoy20.
Area under the concentration versus time curve (AUC) of Decoy20 | Up to 3 years
  The blood pharmacokinetic parameter, AUC, will be assessed pre-dose and up to 28 days post-dose after administration of Decoy20.
Elimination half-life (t1/2) of Decoy20 | Up to 3 years
  The blood pharmacokinetic parameter, t1/2, will be assessed pre-dose and up to 28 days post-dose after administration of Decoy20.
Objective Response Rate (ORR) | Up to 3 years
  ORR is defined as the proportion of subjects achieving a best overall response of confirmed Partial Response (PR) or Complete Response (CR), per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Duration of Response (DoR) | Up to 3 years
  DoR is defined as the duration of time from date of first response to date of disease progression, as per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Indaptus Therapeutics, Study Director — Indaptus Therapeutics, Inc
Locations (12):
- United States (12):
  - University of Southern California- Norris Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - The Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, Siteman Cancer Center, St Louis, Missouri
  - Atlantic Health System, Morristown, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Gabrail Cancer & Research Center, Canton, Ohio
  - UH Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Prisma Health Cancer Institute-ITOR, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newman MJ. Invention and characterization of a systemically administered, attenuated and killed bacteria-based multiple immune receptor agonist for anti-tumor immunotherapy. Front Immunol. 2024 Nov 7;15:1462221. doi: 10.3389/fimmu.2024.1462221. eCollection 2024. PMID 39606250